CLINICAL TRIAL: NCT00967590
Title: A Multi-center, Randomized, Double-Blind, Multiple-Dose, Placebo-controlled Asthma Control Study Evaluating the Efficacy, Safety, and Tolerability of RO5036505 in Subjects With Moderate-to-Severe Asthma
Brief Title: A Study of RO5036505 in Patients With Moderate to Severe Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients dosed
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP22666; 2009-013379-23
Record Dates: First submitted 2009-08-21; First posted 2009-08-28 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO5036505
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RO5036505 — 380mg iv infusion once weekly for 8 weeks
  Arms: 1
Drug: placebo — iv infusion once weekly for 8 weeks
  Arms: 2

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy, safety and tolerability of RO5036505 in patients with inadequately controlled moderate to severe asthma. Patients will be randomized to receive either RO5036505 (380mg iv infusion once weekly) or placebo for 8 weeks. Patients will be on a standardized inhaled corticosteroid/long-acting beta-agonist regimen during study treatment. Target sample size is 50-100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age
* moderate to severe asthma for >/=2 years
* ACQ score >/= 1.5
* ICS and LABA regimen at moderate to high dose
* non-smokers

Exclusion Criteria:

* oral corticosteroid use within 4 weeks prior to screening
* current escalating immunotherapy
* acute infection/antibiotic therapy within 4 weeks prior to screening, or chronic infection
* pulmonary disease other than asthma
* therapy with any approved monoclonal antibody or biologic agent within 12 months prior to screening
* previous exposure to investigational monoclonal antibodies or biologics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
ACQ questionnaire, spirometry assessments, PEFR | every week up to day 95
Safety and tolerability: AEs, spirometry, concomitant medications, laboratory parameters | assessed every week, laboratory parameters every 3-4 weeks, up to day 95

SECONDARY OUTCOMES:
Pharmacokinetics: AUC, Cmax, t1/2, V steady-state, clearance | sampling every week up to day 95

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (14):
  - Little Rock, Arkansas
  - San Diego, California
  - Denver, Colorado
  - Normal, Illinois
  - River Forest, Illinois
  - Boston, Massachusetts
  - St Louis, Missouri
  - Omaha, Nebraska
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Spartanburg, South Carolina
  - Galveston, Texas
  - Madison, Wisconsin
- United Kingdom (2):
  - Hereford
  - Manchester